CLINICAL TRIAL: NCT02801032
Title: The Effect of Tadalafil on Cerebral Large Arteries in Stroke Patients
Brief Title: Effect of Tadalafil on Cerebral Large Arteries in Stroke
Acronym: ETLAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christina Kruuse (Other)
Responsible Party: Sponsor-Investigator, Christina Kruuse, MD, PhD, DMSc, Consultant Neurologist, Associate Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-16020836; 2016-000896-26 (EudraCT Number)
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Stroke, Lacunar; Cerebral Small Vessel Diseases
MeSH Terms: conditions — Stroke, Lacunar; Cerebral Small Vessel Diseases | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Treatment (Active Comparator): Tadalafil 20 mg Capsule. MRI of cerebrum pre dose. Transcranial Doppler, near-infrared spectroscopy (NIRS), endothelial response with EndoPAT2000, and endothelial biomarkers (pre and post dose).
  Interventions: Drug: Tadalafil
- Control (Placebo Comparator): Placebo Capsule. MRI of cerebrum pre dose. Transcranial Doppler, near-infrared spectroscopy (NIRS), endothelial response with EndoPAT2000, and endothelial biomarkers (pre and post dose).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Single dose, 20 mg capsule p.o. minimum one week apart from placebo.
  MRI of cerebrum before the first trial day.
  Transcranial Doppler to measure blood flow velocity in MCA bilaterally before and after intervention.
  Near-infrared spectroscopy (NIRS) to measure cortical brain oxygenation before and after intervention.
  EndoPAT2000 to estimate endothelial function before and after intervention.
  Endothelial biomarkers in blood samples before and after intervention.
  Other Names: Cialis
  Arms: Active Treatment
Drug: Placebo — Single dose, matching capsule p.o. minimum one week apart from active treatment.
  MRI of cerebrum before the first trial day.
  Transcranial Doppler to measure blood flow velocity in MCA bilaterally before and after intervention.
  Near-infrared spectroscopy (NIRS) to measure cortical brain oxygenation before and after intervention.
  EndoPAT2000 to estimate endothelial function before and after intervention.
  Endothelial biomarkers in blood samples before and after intervention.
  Arms: Control

SUMMARY:
In a double blind placebo-controlled cross-over study the effect of tadalafil on blood flow velocity in the large arteries of the brain, cortical brain oxygenation, peripheral endothelial function, and endothelial biomarkers will be tested in patients with lacunar stroke caused by cerebral small vessel disease.

DETAILED DESCRIPTION:
Stroke frequently causes death and decreased function in the everyday life, and the disease has a great human and economic impact. Cerebral small vessel disease (SVD) is the underlying cause of 25 % of all ischemic cerebral strokes and it can further lead to vascular cognitive impairment (VCI), disability and in some cases vascular dementia (VaD). It is well known that cerebral blood flow (CBF) is reduced in VCI. To be able to improve the blood flow in the vasculature of white and gray matter is therefore desirable in slowing the pathology of VCI.

The nitric oxide-cGMP vasodilator pathways has been shown to be impaired in endothelial dysfunction which is seen in SVD.This study targets this well-established mechanism of action by use of a compound selectively inhibiting the breakdown of cGMP, the PDE5 inhibitor tadalafil.

The overall hypothesis is that chronic PDE5 inhibition with tadalafil will lessen the severity and progression of vascular brain lesions via augmentation of cerebral blood flow in the deep brain areas. The specific primary hypothesis for the current project is that PDE5 inhibition with a single dose of tadalafil (Cialis®) will, in contrast to placebo, temporarily change the blood flow in the large blood vessels in the brain and change cortical brain oxygenation in patients with cerebral small vessel disease measured with Transcranial Doppler and near-infrared spectroscopy (NIRS). The secondary hypothesis is that tadalafil will improve the peripheral endothelial function measured as improved blood vessel response in the fingers after a brief occlusion of the arm's blood supply measured with EndoPAT2000. In addition there will be a change of endothelial function biomarkers in the blood after a single dose of tadalafil, and these changes are consistent with the measured peripheral and central blood vessel function.

In regulation of cerebral artery flow and neuronal signalling nitric oxide (NO) and cGMP act as key molecules. In animal models, selective inhibitors of the cGMP degrading PDE5, sildenafil and tadalafil, have been reported to improve the associated symptoms of endothelial dysfunction and stroke recovery. Pre-clinical studies support a CBF-enhancing action of PDE5 inhibitors in cerebrovascular disease while human studies to date have been limited to sildenafil and have not specifically addressed effects on CBF in people with SVD.

Tadalafil (Cialis®; Eli Lilly) is widely prescribed for erectile dysfunction in men. It is also registered for regular daily use at a dose of 40 mg for pulmonary hypertension and 5 mg for benign prostatic hyperplasia. The side effects of tadalafil is well-known and the medicine is usually well tolerated. Tadalafil was chosen over other PDE5 inhibitors (such as sildenafil, Viagra®) due to it's potency, plasma half-life, selectivity for PDE5, and documented brain penetration.

ELIGIBILITY:
Inclusion Criteria:

1. Radiological evidence of cerebral small vessel disease defined as: MRI evidence of lacunar infarct(s) (≤ 1.5 cm maximum diameter) and/or confluent deep white matter leukoaraiosis (≥ grade 2 on Fazekas scale).
2. Clinical evidence of cerebral small vessel disease can be:

   1. lacunar stroke syndrome with symptoms lasting >24 hours occurring at least 5 months previously; OR
   2. transient ischemic attack (TIA) lasting < 24 hours with limb weakness, hemi-sensory loss or dysarthria at least 5 months previously AND with MR DWI performed acutely showing lacunar infarction, OR if MRI is not performed within ten days of TIA, a lacunar infarction in an anatomically appropriate position is demonstrated on a subsequent MRI.
3. Age ≥ 50 years.
4. Imaging of the carotid arteries with Doppler ultrasound, CT angiography, or MR angiography in the previous 12 months demonstrating < 70% stenosis in both internal carotid arteries.

Exclusion Criteria:

1. Known diagnosis of dementia
2. Pregnancy or nursing
3. Cortical infarction (>1.5 cm maximum diameter)
4. Systolic BP < 90 and/or diastolic BP < 50
5. eGFR < 30 ml/min/1,73m2
6. Severe hepatic impairment
7. History of Lactose intolerance
8. Concomitant use of PDE5 inhibitors e.g. sildenafil, tadalafil, vardenafil
9. Patients receiving nicorandil and nitrates e.g. isosorbide mononitrate, isosorbide dinitrate, glyceryl trinitrate
10. Body weight > 130kg
11. Uncontrolled cardiac failure
12. Persistent or paroxysmal atrial fibrillation
13. History of "sick sinus syndrome" or other supraventricular cardiac conduction conditions such as sinoatrial or atrioventricular block
14. Uncontrolled COPD
15. Stroke or TIA within the last 5 months.
16. MRI not tolerated or contraindicated: MRI exclusion criteria: Participant has a cardiac pacemaker; recent surgery; vascular clips; metal implants or joint replacements that are not compatible with MRI; have had metal fragments in their eyes; has ever worked on a lathe; has shrapnel from a war injury; possibility of pregnancy
17. Known monogenic causes of stroke i.e. CADASIL
18. The patient does not wish to know important results from MRI
19. Unable to provide informed consent
20. Not possible to localise a. cerebri media bilaterally on inclusion day with Transcranial Doppler

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
Difference in Blood flow velocity change in middel cerebral artery (MCA) between placebo and tadalafil | Measurement before and up to three hours after intake of tadalafil/placebo.
  Change in Blood flow velocity in middel cerebral artery (MCA) will be measured with transcranial doppler (TCD) before and up to three hours after intake of tadalafil/placebo.
Difference in cortical brain oxygenation between placebo and tadalafil | Measurement before and up to three hours after intake of tadalafil/placebo.
  Cortical brain oxygenation will be measured with near-infrared spectroscopy (NIRS) before and up to three hours after intake of tadalafil/placebo.

SECONDARY OUTCOMES:
Changes in endothelial response | Measurement before and three hours after intake of tadalafil/placebo.
  Measurement of endothelial response by EndoPAT2000 before and three hours after intake of tadalafil/placebo.
Changes in endothelial biomarkers in blood | Blood samples before and 3,5-4 hours after intake of tadalafil/placebo.
  Blood samples to measure changes in endothelial biomarkers (eg. e-selectin, VCAM, ICAM, endothelin, ADMA, miRNA) before and 3,5-4 hours after intake of tadalafil/placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Christina R Kruuse, MD, PhD, Principal Investigator — Consultant Neurologist, Dept Neurology, Herlev Hospital
Locations (1):
- Department of Neurology, Herlev-Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No